CLINICAL TRIAL: NCT01322841
Title: Universal Screening for Tuberculosis and Anemia With the CHICA System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Principal Investigator, Aaron Carroll, Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CHICA_Screening; 5K22LM009160 (NIH)
Record Dates: First submitted 2011-03-23; First posted 2011-03-25 (Estimated); Results first posted 2015-12-18 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-10

CONDITIONS: Tuberculosis; Iron Deficiency Anemia
Keywords: CHICA; clinical decision support
MeSH Terms: conditions — Tuberculosis; Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHICA Diagnosis Module (Active Comparator): This arm had the CHICA screening module turned on
  Interventions: Other: CHICA Diagnosis Module
- CHICA Placebo (Placebo Comparator): This arm had CHICA but no additional module
  Interventions: Other: CHICA Placebo

INTERVENTIONS:
Other: CHICA Diagnosis Module — The CHICA module helped to screen and diagnose patients with tuberculosis or iron deficiency anemia
  Arms: CHICA Diagnosis Module
Other: CHICA Placebo — This was CHICA without the screening module
  Arms: CHICA Placebo

SUMMARY:
The CHICA system is a clinical decision support system that uses adaptive turnaround documents to provide point-of-care information to clinicians. The investigators will be studying whether it can help in the diagnosis and treatment of tuberculosis and iron deficiency anemia.

DETAILED DESCRIPTION:
The CHICA system is a clinical decision support system that uses adaptive turnaround documents to provide point-of-care information to clinicians. We will be studying whether it can help in the diagnosis and treatment of tuberculosis and iron deficiency anemia.

ELIGIBILITY:
Inclusion Criteria:

Age 3 to 11 years old and seen in a study clinic

Exclusion Criteria:

None

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2239 (Actual)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron E Carroll, MD, MS, Principal Investigator — IUSM
Locations (1):
- Children's Health Services Research, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- CHICA Diagnosis Module: This arm had the CHICA screening module turned on CHICA diagnosis module: The CHICA module helped to screen and diagnose patients with tuberculosis or iron deficiency anemia
- CHICA Placebo: This arm had CHICA but no additional module CHICA Placebo: This was CHICA without the screening module
Period: Overall Study
Arm/Group | CHICA Diagnosis Module | CHICA Placebo
Started | 1116 | 1123
Completed | 1116 | 1123
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHICA Diagnosis Module | CHICA Placebo | Total
Number analyzed (Participants) | 1116 | 1123 | 2239
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1116 | 1123 | 2239
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 538 | 542 | 1080
  Male | 578 | 581 | 1159
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 21 | 27 | 48
  Black or African American | 394 | 397 | 791
  White | 679 | 662 | 1341
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 20 | 37 | 57

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Screened Positive for One of the Disorders
Time Frame: six months
Measure: Number; unit: percentage of participants
Arm/Group | CHICA Diagnosis Module | CHICA Placebo
Number analyzed (Participants) | 1116 | 1123
percentage of participants
  Iron Deficiency | 17.5 | 3.1
  TB | 1.8 | 0.8

2. Secondary Outcome: Percentage of Patients Diagnosed With One of the Disorders
Time Frame: six months
Measure: Number; unit: percentage of participants
Arm/Group | CHICA Diagnosis Module | CHICA Placebo
Number analyzed (Participants) | 1116 | 1123
percentage of participants
  Iron Deficiency Anemia | 0.3 | 0
  TB | 0.2 | 0

ADVERSE EVENTS:
Time Frame: six months
Arm/Group | CHICA Diagnosis Module | CHICA Placebo
Serious Adverse Events (participants affected / at risk) | 0/1116 | 0/1123
Other Adverse Events (participants affected / at risk) | 0/1116 | 0/1123

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No